CLINICAL TRIAL: NCT01998204
Title: Requirement of Propofol for Induction of Unconsciousness in Patients With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Jia-feng Wang, Dr., Changhai Hospital
Other Study IDs: Parkinson-propofol
Record Dates: First submitted 2013-11-19; First posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; propofol; deep brain stimulator
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PD group: Patients with Parkinson's disease undergoing deep brain stimulator implantation and pulse generator placement
- non-PD group: Patients without Parkinson's disease undergoing intracranial surgery

SUMMARY:
Parkinson's disease (PD) is the second most prevalent neurodegenerative disease. The investigators clinical experience showed a trend of delayed emergence among patients undergoing deep brain stimulator (DBS) implantation and pulse generator placement under general anesthesia. Abnormal pharmacodynamics might be present among these patients, which had never been investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's disease undergoing deep brain stimulator implantation and pulse generator placement under general anesthesia
* non-Parkinsonian patients without Parkinson's disease undergoing intracranial surgery under general anesthesia

Exclusion Criteria:

* ASA score higher than Class III
* predicted difficult airway
* hearing impairment
* inability to corporate with instruction
* alcohol or drug abuser
* patients refusing to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study recruits patients with Parkinson's disease undergoing deep brain stimulator implantation and pulse generator placement under general anesthesia and non-Parkinsonian patients without Parkinson's disease undergoing intracranial surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Consciousness status | Participants will be monitored during the period of propofol infusion, an expected average of less than 10 min
  Consciousness status is evaluated by the observer's assessment of alertness and sedation score (OAA/S).

CONTACTS AND LOCATIONS:
Overall Officials: Jia-feng Wang, M.D., Principal Investigator — Department of Anesthesiology, Changhai Hospital, Second Military Medical University
Locations (1):
- Department of Anesthesiology, Changhai Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Xu XP, Yu XY, Wu X, Hu XW, Chen JC, Li JB, Wang JF, Deng XM. Propofol requirement for induction of unconsciousness is reduced in patients with Parkinson's disease: a case control study. Biomed Res Int. 2015;2015:953729. doi: 10.1155/2015/953729. Epub 2015 Oct 1. PMID 26495319